CLINICAL TRIAL: NCT01339715
Title: From the Changes of Ryodoraku Value at 12 Source Acupoints, and Heart Rate Viability to Explain the Difference Between Acupuncture and Far-infrared Ray Illumination at CV12（Zhongwan）Acupoint
Brief Title: The Difference Between Acupuncture and Far-infrared Ray Illumination at CV12 Acupoint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DMR100-IRB-032
Record Dates: First submitted 2011-04-17; First posted 2011-04-21 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Reaction of Autonomic Nervous System; Reaction of Acupuncture; Reaction of Far Infrared Ray
Keywords: Ryodoraku; Heart Rate Variability; Traditional medicine; Autonomic Nervous System; Acupuncture; Far Infrared Ray; CV12 Acupoint
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: acupuncture and far-infrared ray — During experimental phase,inserting the needle of acupuncture into CV12 acupoint or using far-infrared ray to illuminate on CV12 20 minutes.

SUMMARY:
The purpose of the study was to investigate the changes of Ryodoraku value at 12 source acupoints, and heart rate viability (HRV) when acupuncture or far-infrared ray illumination applied to CV12 acupoint.

DETAILED DESCRIPTION:
Acupuncture and far-infrared ray illumination at CV12 acupoint have been widely used to treat many diseases in clinic. To our knowledge, the report is about the different reaction on autonomic nervous system between acupuncture and far-infrared illumination is very rare until now.Therefore,the study was to investigate the different changes on autonomic nervous system from Ryodoraku value at 12 source acupoints and heart rate viability (HRV) when acupuncture or far-infrared ray illumination applied to CV12 acupoint.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, male or female, ages between 20 and 40
* Neurological and physical examination without abnormal functions
* Far-infrared ray illumination without allergic reaction and contra- indication
* The participants were explained the objective of the study, agreed to accept the test and signed a letter of consent

Exclusion Criteria:

* People less than 20 years of age or more than 40 years
* Women in pregnant or lactating
* People with mental or behavioral anomalies could not follow the researchers
* People with pacemakers
* People suffered from serious diseases such as myocardial infarction , heart failure, serious arrhythmia, hypertension, diabetes, autoimmune disease, chronic obstructive pulmonary diseases, and kidney failure, liver cirrhosis and cancer
* People accepted acupuncture and moxibustion in a week, or were taking any drugs for treatment
* People suffered from limb edema and serious skin diseases
* People with excessive obesity (body mass index, BMI>30)
* People did not sign a letter of consent

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
From the changes of Ryodoraku value at 12 source acupoints, and heart rate viability to measure the difference | Each period was 20 min in duration. The Ryodoraku value of 12 source acupoints were measured, and 5-min HRV was recorded at the end of each period.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, professor, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan